CLINICAL TRIAL: NCT01926756
Title: Intraoperative One-Time Catheterization in Short Gynecologic Procedures and Its Potential Effect on Symptomatic and Asymptomatic Bacteriuria
Brief Title: Does Straight Catheterization in Short Gynecologic Procedures Cause Bacteriuria?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abington Memorial Hospital (Other)
Responsible Party: Principal Investigator, Emily G. Parent, D.O., OB/GYN Resident Physician PGY-IV, Abington Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AMH-Myers/Parent001
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Postoperative Bacteriuria
Keywords: bacteriuria; straight catheterization; urinary tract infections; iatrogenic
MeSH Terms: conditions — Bacteriuria; Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Straight catheterization (control) (Other): The control arm is the current practice at our hospital (to perform straight catheterization for short procedures).
  Interventions: Procedure: Straight catheterization
- No straight catheterization (Active Comparator): The experimental arm will void preoperatively and will not be straight catheterized intraoperatively. This is a change from the current practice at our hospital.
  Interventions: Procedure: No straight catheterization

INTERVENTIONS:
Procedure: Straight catheterization — Patient will receive the current standard practice of straight catheterization intraoperatively.
  Arms: Straight catheterization (control)
Procedure: No straight catheterization — Patients will not be catheterized which is an experimental change from the current practice at our hospital.
  Arms: No straight catheterization

SUMMARY:
This is a prospective randomized controlled trial to look into the reduction of catheter associated urinary tract infections in the postoperative period. It will specifically look at short gynecologic procedures such as D&C (dilation and curettage), hysteroscopies and LEEP procedures and the need to perform intraoperative catheterization. If a patient urinates immediately before a short operation then there is no need to drain the bladder with a catheter during the procedure. The investigators hypothesize that eliminating catheterization during these short procedures may decrease postoperative urinary tract infections. The hope is that this study would provide evidence to support a change in practice.

DETAILED DESCRIPTION:
The majority of research currently concentrates on indwelling catheters rather than one-time catheterization. Current practice at our institution in the gynecologic operating room is to perform a one time catheterization on patient's undergoing short procedures, yet it is unclear if this is a necessary intervention. If patients are asked to void immediately before their procedure it would eliminate the need for intra-operative catheterization and eliminate a potential source of infection.

The study is designed to determine whether routine catheterization prior to a minor OB/GYN procedure causes symptomatic or asymptomatic bacteria in the urine. Current practice is one-time catheterization of patients undergoing minor OB/GYN procedures prior to the beginning of the procedure. The investigators hypothesize that this causes asymptomatic or symptomatic bacteriuria.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be 18 years of age or older.
* The patient must be female.
* The patient must be undergoing a same-day gynecologic procedure where catheterization is usually performed.
* The patient must have general anesthesia or monitored anesthesia care (MAC). This includes IV sedation.

Exclusion Criteria:

* The patient cannot be undergoing intermittent one-time catheterization.
* The patient can not have had an indwelling catheter placed in the past 6 months.
* The patients cannot have a concomitant pelvic infection.
* The procedure cannot require spinal anesthesia.
* The patient cannot be taking immunosuppressive medications.
* The patient cannot be taking antibiotics and/or suppressive therapy for chronic urinary tract infections.
* The patient cannot receive pre-operative or intra-operative antibiotics.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative Bacteriuria | 2 -4 weeks
  Urine cultures are obtained preoperatively (baseline), immediately postoperatively and 2 to 4 weeks postoperatively.

SECONDARY OUTCOMES:
Subjective urinary tract discomfort | 2-4 weeks postoperatively

OTHER OUTCOMES:
Symptomatic urinary tract infection | 2-4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Emily G Parent, D.O., Principal Investigator — Abington Memorial Hospital
Locations (1):
- Abington Memorial Hospital, Abington, Pennsylvania, United States